CLINICAL TRIAL: NCT04666701
Title: National, Multicenter, Randomized, Double-blind, Triple-dummy, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Escócia Association in the Treatment of Acute Pain
Brief Title: Efficacy and Safety of Escócia Association in the Treatment of Acute Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategy review
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS1319 - ESCÓCIA
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Ketorolac Tromethamine; Scopolamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Escócia association (Experimental): The study is triple-dummy. The patient must take 3 pills, with a minimum interval of 6/6 hours for a maximum of 5 days, if pain, as follows:
  1 tablet Escócia association, oral
  1 dragee Placebo Scopolamine, oral
  1 tablet Placebo Ketorolac, sublingual
  Interventions: Drug: Escócia association; Other: Placebo Ketorolac; Other: Placebo Scopolamine
- Ketorolac (Active Comparator): The study is triple-dummy. The patient must take 3 pills, with a minimum interval of 6/6 hours for a maximum of 5 days, if pain, as follows:
  1 tablet Ketorolac, sublingual
  1 tablet Placebo Escócia association, oral
  1 dragee Placebo Scopolamine, oral
  Interventions: Other: Placebo Scopolamine; Drug: Ketorolac Tromethamine; Other: Placebo Escócia association
- Scopolamine (Active Comparator): The study is triple-dummy. The patient must take 3 pills, with a minimum interval of 6/6 hours for a maximum of 5 days, if pain, as follows:
  1 dragee Scopolamine, oral
  1 tablet Placebo Ketorolac, sublingual
  1 tablet Placebo Escócia association, oral
  Interventions: Other: Placebo Ketorolac; Drug: Scopolamine; Other: Placebo Escócia association

INTERVENTIONS:
Drug: Escócia association — Escócia association tablet
  Arms: Escócia association
Other: Placebo Ketorolac — Placebo Ketorolac tablet
  Arms: Escócia association; Scopolamine
Other: Placebo Scopolamine — Placebo Scopolamine dragee
  Arms: Escócia association; Ketorolac
Drug: Ketorolac Tromethamine — Ketorolac tablet
  Arms: Ketorolac
Drug: Scopolamine — Scopolamine dragee
  Arms: Scopolamine
Other: Placebo Escócia association — Placebo Escócia association tablet
  Arms: Ketorolac; Scopolamine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Escócia association in adults with acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Participants, aged 18 years and older, with renal colic admitted in the emergency service, or those who underwent an extracorporeal lithotripsy procedure to eliminate kidney stones.

Exclusion Criteria:

* Known hypersensitivity to the formula components used during the clinical trial;
* History of alcohol and/or substance abuse within 2 years;
* Pregnant women, breastfeeding or planning to become pregnant, or women with the potential to become pregnant who are not using a reliable method of contraception;
* Participants weighing less than 50 kg;
* Participants with suspected other causes of acute abdominal pain;
* Participants with a known history of peptic ulcer, gastrointestinal bleeding, perforation or inflammatory bowel disease;
* Participants with hypovolemia or dehydration;
* Renal failure, defined by the estimated glomerular filtration rate [eGFR] <60 mL / min / 1.73 m2;
* Participants with a known medical history of cerebrovascular bleeding, hemorrhagic diathesis (hemophilia), blood clotting disorders; postoperative of coronary artery bypass graft surgery, or using anticoagulants, including low heparin dose (2500-5000 units every 12 hours);
* Participants in the postoperative period with a high risk of bleeding or incomplete homeostasis;
* Participants with cardiovascular disease, chronic heart failure or with increased risk of cardiovascular events are at the discretion of the investigator, in order to include the participant;
* Participants with a current medical history of cancer and / or cancer treatment in the last 5 years;
* Participants using pentoxifylline, probenecid or lithium salts;
* Participants with megacolon and / or paralytic or obstructive ileus;
* Participants with glaucoma and myasthenia gravis;
* Participants on treatment with MAO inhibitors, or participants who have been treated with these drugs within 14 days;
* Participants on epilepsy not adequately controlled treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain intensity | 0-1 hour
  The change from baseline in pain intensity 1 hour after using the first dose of medication. Pain intensity will be assessed by visual analog scale (VAS), between 0 cm (no pain) and 10 cm (worst pain), recorded in the participant's diary.

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study | 10 days
  Incidence and severity of adverse events recorded during the study over 10 days.

IPD SHARING:
Plan to Share IPD: No